CLINICAL TRIAL: NCT05551351
Title: CT av förkalkade kranskärl Med fotonräknarteknik
Brief Title: CT in Calcified Coronary Arteries With Photon Counting Detector
Acronym: CCT-PCD-1
Status: Terminated | Type: Observational
Why Stopped: Enrollment rate too slow to reach anticipated number of participants.
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: 278326
Record Dates: First submitted 2022-09-13; First posted 2022-09-22 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Coronary Stenosis; Calcific Coronary Arteriosclerosis
Keywords: Cardiac Computed Tomography; Photon Counting Detector
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Coronary CT: The single cohort consists of all patients enrolled in the study. All participants performs cardiac CT and coronary angiography as part of routine care.
  Interventions: Diagnostic Test: Cardiac CT with photon counting detector

INTERVENTIONS:
Diagnostic Test: Cardiac CT with photon counting detector — Cardiac CT including the coronary arteries. The cardiac CT is performed in routine care for the included patients.

SUMMARY:
Coronary CT angiography is challenging in patients with more than mildly calcified coronary vessels, because of calcium artefacts that prevents evaluation of the lumen. The purpose of the CCT-PCD-1-study is to evaluate the diagnostic accuracy and image quality in coronary CT angiography using a commercially available CT system equipped with a photon counting detector technology.

Patients referred for cardiac CT and conventional coronary angiography as part of routine preoperative evaluation before Transcatheter Aortic Valve Implantation (TAVI) will be asked for inclusion in the study. This group of patients has generally a coronary artery calcium burden and perform cardiac CT and coronary angiography as part of routine care.

The diagnostic accuracy concerning significant coronary artery stenosis on the preoperative CT will be evaluated with the conventional coronary angiography as reference. Also, CT examination image quality will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for cardiac CT AND conventional coronary angiography as part of routine preoperative evaluation.

Exclusion Criteria:

* <65 years old.
* Heart arrhythmia.
* Heart rate >90/min with contraindication against beta blockers.
* Not capable of giving informed consent
* eGFR <30 mL/min/1.73m2

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population are at least 65 years old with an expected median age of ~80 years. This group of patients has generally a high coronary artery calcium burden which prevents conventional cardiac CT from evaluation of the coronary arteries.
  Since cardiac CT and coronary artery angiography is performed as part of routine care in this patient cohort, no extra examinations are needed for the reference measure of the primary outcome.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of CT concerning coronary stenosis with conventional angiography as reference | 1 day. (Coronary angiography is usually performed the same day as cardiac CT.)
  Coronary angiography with or without FFR is performed as part of routine care for included patients. The outcome measure is the agreement between coronary CT and coronary angiography.

SECONDARY OUTCOMES:
Image quality | 1 day. (Image quality is assessed on the performed examination)
  Image quality on CT examination according to European guidelines on quality criteria for computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Mats Lidén, MD, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Röntgenkliniken Universitetssjukhuset Örebro, Örebro, Sweden